CLINICAL TRIAL: NCT00893607
Title: Proof of Concept Study in Healthy Volunteers to Investigate the Safety and Response to a Single Dose of 10mg Methoxamine (NRL001) Applied Locally Using a Suppository to the Anal Canal or Rectum
Brief Title: Effect of Single Doses of 10 mg NRL001 Applied as a Suppository to the Anal Canal or Rectum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Hans-Jürgen Gruss, Norgine Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRL001-01/2006 (SUPP)
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-anal (Experimental): The first 12 subjects were administered 10mg NRL001 as a slow release suppository into the anal canal.
  Interventions: Drug: NRL001
- Rectal (Experimental): The second 12 subjects were administered 10mg NRL001 as a slow release rectal suppository.
  Interventions: Drug: NRL001

INTERVENTIONS:
Drug: NRL001 — 10mg NRL001 was administered as a slow release suppository
  Other Names: Methoxamine Hydochloride

SUMMARY:
Study to assess the effects of 10mg NRL001 on mean anal resting pressure (MARP) when administered as a slow release suppository applied to the anal canal or rectum. In addition, the pharmacokinetics of NRL001 in plasma, adverse events, and any changes in heart rate or blood pressure were to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* No previous history of ano-rectal conditions/ diseases
* No history of cardiovascular disease
* 18 to 75 years of age
* Males and females (pre-menopausal females of child-bearing potential must be using adequate contraceptive methods and have a negative pregnancy test before the start of the study)

Exclusion Criteria:

* Use of medication in the last 30 days with a vasodilatory activity
* Use of monoamine oxidase inhibitors (MAOI) presently or within the last two weeks before study participation
* Use of any medication in the last 30 days applied to the anus and/or via the rectum (exception: participation in NRL001-01/2006 (SUPP) for previous dosing into the anal canal)
* Application of any unlicensed medication within the previous 3 months (exception: participation in NRL001-01/2006 (SUPP))
* Regular intake of more than 21 units of alcohol per week
* History or any evidence of cardiovascular disease including ischaemic heart disease and hypertension (defined on examination: systolic blood pressure greater than 160mmHg or diastolic blood pressure greater than 90mmHg; based on at least two separate readings), peripheral vascular disease or Raynaud's syndrome
* Presence of diabetes mellitus
* History or symptoms of thyroid diseases, including hypo- or hyperthyroidism
* Pregnant females
* Breast feeding mothers
* Presence of concomitant gastrointestinal diseases or disorders, such as significant abdominal symptoms and haemorrhoids but also any significant organ (e.g. renal, hepatic or cardiac) dysfunction
* Volunteers whom the investigator feels would not be compliant with the requirements of the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in mean anal resting pressure (MARP) | Up to 6 hours post-dose

SECONDARY OUTCOMES:
Pharmacokinetics of NRL001 in plasma | Up to 6 hours post-dose
Monitoring of blood pressure and heart rate | Up to 6 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: John H Scholefield, Principal Investigator — University Hospital - Queens Medical Centre
Locations (1):
- Division of GI Surgery, University Hospital - Queens Medical Centre, Nottingham, United Kingdom